CLINICAL TRIAL: NCT04564586
Title: Developing and Testing a Technology-Based Translation of the Diabetes Prevention Program for Adult Primary Care Patients At-Risk of Developing Type 2 Diabetes Mellitus
Brief Title: Developing and Testing a Technology-Based Translation of the DPP to Address Prediabetes in a Primary Care Setting
Acronym: DPPFit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Jessica Lynn Stewart, PhD, MPH, Principle Investigator, Augusta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB#1193356
Record Dates: First submitted 2020-08-27; First posted 2020-09-25 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: PreDiabetes; Metabolic Syndrome, Protection Against
Keywords: mHealth; real-world setting; primary care intervention; diabetes prevention; remote; translation
MeSH Terms: conditions — Prediabetic State; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enhanced Intervention Group (EIG) (Other): The Enhanced Intervention Group was a subgroup of the participants that were invited for voluntary weekly meet-n-greet sessions in the Primary Care Clinic. These sessions were information and not educational sessions for the intervention. The entire EIG concept was to test a social component of participants by providing an informal opportunity for a DPPFit social group. The group sessions were terminated after only 5 weeks as a result of the Covid-19 pandemic. They were the only component of the DPPFit study that were face-to-face.
  Interventions: Behavioral: DPPFit

INTERVENTIONS:
Behavioral: DPPFit — Participants issued Fitbit Device and set up Fitbit App. They are then enrolled in the automated text messaging platform. Day 1 of the intervention begins the Monday after consent. All consented participants receive the full intervention.

SUMMARY:
DPPFit is a Healthy Lifestyle Intervention designed to reformat the effective strategies of the Diabetes Prevention Program (NDPP) into a tool for use in a primary care setting. DPPFit is a 16-week technology-based intervention for diabetes prevention. In keeping with the National DPP educational sessions, the intervention weeks follow the order and presentation of the N-DPP 16 session topics. The goal is to develop a pragmatic translation of the DPP that is effective in the real-world setting of primary care clinic. The hope is that in doing so, those at risk of developing type II diabetes mellitus will have evidenced-based prevention methods at their disposal.

DETAILED DESCRIPTION:
DPPFit is an HLI designed to translate the effective strategies of the National Diabetes Prevention Program (N-DPP) into a tool for use in a primary care setting. The 16-week intervention follows the order of the 16 sessions that make up the core components of the traditional DPP. The novelty in this application is the intervention delivery, in addition to the use of technology to supplement resource and time intensive DPP behavioral strategies. The entire intervention is delivered through automated text messages (SMS/MMS). For any given week, the daily text messages for that week reflect the core session of the DPP (i.e DPPFit Week 1 texts correspond to DPP Session 1). In addition to the automated daily messages, participants are issued a Fitbit and assisted in setting up the Fitbit App on their smart phones. The Fitbit App is considered a standalone mHealth App. The fitness tracker and companion App allow participants to set goals and track food and physical activity. The content of the text messaging is almost entirely from the N-DPP participant notebook (2012). Exceptions to this are a series of prompts to cue participant to use the Fitbit and/or Fitbit App to support the session. These include topics about setting goals in the Fitbit App, how to track food using the App, or how to connect with friends and do challenges on Fitbit.

To be sustainable and feasible in a primary care setting, remote delivery of intervention materials and components is a necessary part of any evidence-based tool to address diabetes prevention. This automated, remote dissemination, technology-based application of the N-DPP components means that intervention delivery and protocol are feasible methods to address diabetes prevention in light of the ongoing Covid-19 health crisis.

ELIGIBILITY:
Inclusion Criteria:

* Non-institutionalized adult patients
* Ages 18 - 55 years
* Diagnosed as prediabetes or with HbA1c% values between 5.7-6.4%.

Exclusion Criteria:

* Prior bariatric surgery
* Participation in weight loss program or current weight loss medication.
* History of T1DM or T2DM diagnosis
* Use of medications to treat glucose intolerance, including biguanides and sulfonylureas.
* History of infarction, angina, coronary artery bypass graft surgery, coronary angioplasty, congestive heart failure, or any condition that significantly limits their exercise such as peripheral arterial disease.
* BMI (kg/m²)< 18.5

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 12 Months
  Weight Loss by % of change and total weight change (kg)
Physical Activity | 6 months
  Physical activity days/week, change > 10% of PA, Kcal/week
Inactivity | 6 months
  Change in Sedentary Time, Mins/day

SECONDARY OUTCOMES:
Health Related Quality of Life | 6 months
  MOS SF-20 / MOS Social Support Scale
Hemoglobin A1c | 12 months
  Change in % of HbA1c at 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Stewart, MPH, Principal Investigator — Augusta University
Locations (1):
- Augusta University - General Internal Medicine Clinic, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coughlin SS, Stewart J. Use of Consumer Wearable Devices to Promote Physical Activity: A Review of Health Intervention Studies. J Environ Health Sci. 2016 Nov;2(6):10.15436/2378-6841.16.1123. doi: 10.15436/2378-6841.16.1123. Epub 2016 Nov 30. PMID 28428979